CLINICAL TRIAL: NCT01555684
Title: The Effect of Percutaneous Venoplasty on Muscular Function, Mobility and Fatigue of Multiple Sclerosis (MS) Patients With Chronic Cerebrospinal Venous Insufficiency (CCSVI).
Brief Title: Functional Changes Following Percutaneous Venoplasty in Multiple Sclerosis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Dr Angus Hunter, Principal Investigator, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPREC#501
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis; Chronic Cerebrospinal Venous Insufficiency
Keywords: MS; CCSVI
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- venoplasty proceedures (Experimental): Half of the participants receive treatment and the other half do not
  Interventions: Procedure: percutaneous venoplasty to alleviate chronic cerebrospinal venous insufficiency
- Control - no treatment (Placebo Comparator)
  Interventions: Procedure: percutaneous venoplasty to alleviate chronic cerebrospinal venous insufficiency

INTERVENTIONS:
Procedure: percutaneous venoplasty to alleviate chronic cerebrospinal venous insufficiency — percutaneous venoplasty is where a balloon is inserted and inflated into the jugular vein has been developed to improve this drainage of the CNS, reduce venous hypertension and improve symptoms associated with MS

SUMMARY:
Multiple Sclerosis (MS) is a demyelinating disease of the central nervous system (CNS) that often results in reduced muscle function which produces fatigue, weakness and a decline in daily mobility. Although the underlying cause of the disease is unknown a possible contributory mechanism is chronic cerebrospinal venous insufficiency (CCSVI). Post-mortem studies and magnetic resonance venography have shown a strong relationship between the cerebral venous system and MS cortical plaques. From this a role for CCSVI in MS has been suggested: venous malformations that result in venous hypertension, pressure on the blood brain barrier and subsequent inflammation due to leakage of haemosiderin into the parenchyma. This provokes an immune response which results in neurodegeneration. A procedure known as percutaneous venoplasty whereupon a balloon is inserted and inflated into the jugular vein has been developed to improve this drainage of the CNS, reduce venous hypertension and improve symptoms associated with MS. Although this procedure is widely practiced throughout the world it has yet to be fully accepted as it needs to be supported by evidence based clinical trials. As such NHS National Institute for Health and Clinical Excellence (NICE) recently issued a consultation document to determine more about the procedure's clinical safety and efficacy. A common concern raised is the ability to prevent any possible placebo effect and like any other clinical trial should offer a sham procedure to a matched control group. The difficulty with this option are the ethical issues associated with an invasive sham treatment and also the practical issues of masking a potentially painful treatment such as venoplasty. One option is to have blinded neurological assessment of patients who have either been treated with venoplasty or had no active treatment. Another option is to use dependent measures that are unaffected by motivational or psychological influences which avoids any placebo effect issue. One such dependent measure is motor unit firing behaviour whilst contracting at a submaximal target force. Typically clinicians have used this to manage motor disorder patients but have used cumbersome invasive technology that can only measure a few motor units with limited accuracy. However, De Luca et al recently developed a high density surface electromyographic (HDsEMG) system that can measure 30-40 motor units with 92-97% accuracy. From this it has been proposed as a highly effective tool for evaluating efficacy of therapeutic interventions for upper motoneuron disorders such as MS.

Accordingly the investigators propose to use a repeated measures design on an experimental (receiving venoplasty) and control (not receiving venoplasty) MS groups (6 patients in each group) to determine the effect of the treatment on muscular function, mobility and fatigue. This would be combined with independent blinded neurological assessment of the two groups of patients.

This design enables us to achieve two aims:

1. Acute neuromuscular response to the treatment
2. Chronic response to the treatment (6 weeks) to determine the effect on muscular function, mobility and fatigue.*

Methods

* Four (first two to establish baseline variability of measures) repeat visits to the laboratory at University of Stirling to establish neuromuscular measures:

  1. HDsEMG pre and post tetanic induced fatigue
  2. Muscle fibre conduction velocity as previously described (Hunter et al., 2011)
  3. Ultrasound for CCSVI determination on visits 1 and 3
  4. DEXA scans for alterations in body composition on visits 2 and 4
* With the use of accelerometers monitor free living activity on days 0-7 and 9-42 (post venoplasty).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CCSVI using transcranial and extracranial colour Doppler sonography in both supine and sitting positions. The diagnosis requires that 2 or more of the following 5 criteria are met:

  * reflux in the internal jugular or vertebral veins, or both, with the head in any position
  * reflux in the deep cerebral veins
  * high-resolution B-mode evidence of internal jugular vein stenosis
  * absence of Doppler-detectable flow in the internal jugular veins and/or vertebral veins
  * loss of postural control of the main cerebral venous outflow pathways.

Exclusion Criteria:

* non ambulatory

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular function | 52 days
  The venoplasty procedure will be performed at 8 days

SECONDARY OUTCOMES:
Free living activity | 0-7 and 9-52 days
  Measured by accelerometery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Stirling, Stirling, United Kingdom

REFERENCES:
- [Background] De Luca CJ, Hostage EC. Relationship between firing rate and recruitment threshold of motoneurons in voluntary isometric contractions. J Neurophysiol. 2010 Aug;104(2):1034-46. doi: 10.1152/jn.01018.2009. Epub 2010 Jun 16. PMID 20554838
- [Background] Fog T. The topography of plaques in multiple sclerosis with special reference to cerebral plaques. Acta Neurol Scand Suppl. 1965;15:1-161. No abstract available. PMID 5213727
- [Background] Fox RJ, Rae-Grant A. Chronic cerebrospinal venous insufficiency: have we found the cause and cure of MS? Neurology. 2011 Jul 12;77(2):98-100. doi: 10.1212/WNL.0b013e318212a915. Epub 2011 Apr 13. No abstract available. PMID 21490321
- [Background] Ge Y, Zohrabian VM, Grossman RI. Seven-Tesla magnetic resonance imaging: new vision of microvascular abnormalities in multiple sclerosis. Arch Neurol. 2008 Jun;65(6):812-6. doi: 10.1001/archneur.65.6.812. PMID 18541803
- [Background] Hunter A, Albertus-Kajee Y, St Clair Gibson A. The effect of exercise induced hyperthermia on muscle fibre conduction velocity during sustained isometric contraction. J Electromyogr Kinesiol. 2011 Oct;21(5):834-40. doi: 10.1016/j.jelekin.2011.06.002. Epub 2011 Jul 13. PMID 21745750
- [Background] Kermode AG, Thompson AJ, Tofts P, MacManus DG, Kendall BE, Kingsley DP, Moseley IF, Rudge P, McDonald WI. Breakdown of the blood-brain barrier precedes symptoms and other MRI signs of new lesions in multiple sclerosis. Pathogenetic and clinical implications. Brain. 1990 Oct;113 ( Pt 5):1477-89. doi: 10.1093/brain/113.5.1477. PMID 2245307
- [Background] Kidd D, Barkhof F, McConnell R, Algra PR, Allen IV, Revesz T. Cortical lesions in multiple sclerosis. Brain. 1999 Jan;122 ( Pt 1):17-26. doi: 10.1093/brain/122.1.17. PMID 10050891
- [Background] Nawab SH, Chang SS, De Luca CJ. High-yield decomposition of surface EMG signals. Clin Neurophysiol. 2010 Oct;121(10):1602-15. doi: 10.1016/j.clinph.2009.11.092. Epub 2010 Apr 28. PMID 20430694
- [Background] Tan IL, van Schijndel RA, Pouwels PJ, van Walderveen MA, Reichenbach JR, Manoliu RA, Barkhof F. MR venography of multiple sclerosis. AJNR Am J Neuroradiol. 2000 Jun-Jul;21(6):1039-42. PMID 10871010
- [Background] Imperial College CCSVI Investigation Group; Thapar A, Lane TR, Pandey V, Shalhoub J, Malik O, Ellis M, Franklin IJ, Nicholas R, Davies AH. Internal jugular thrombosis post venoplasty for chronic cerebrospinal venous insufficiency. Phlebology. 2011 Sep;26(6):254-6. doi: 10.1258/phleb.2011.011052. Epub 2011 Jul 29. PMID 21803799
- [Background] Zamboni P, Galeotti R, Menegatti E, Malagoni AM, Tacconi G, Dall'Ara S, Bartolomei I, Salvi F. Chronic cerebrospinal venous insufficiency in patients with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):392-9. doi: 10.1136/jnnp.2008.157164. Epub 2008 Dec 5. PMID 19060024
- [Background] Zamboni P, Menegatti E, Weinstock-Guttman B, Dwyer MG, Schirda CV, Malagoni AM, Hojnacki D, Kennedy C, Carl E, Bergsland N, Magnano C, Bartolomei I, Salvi F, Zivadinov R. Hypoperfusion of brain parenchyma is associated with the severity of chronic cerebrospinal venous insufficiency in patients with multiple sclerosis: a cross-sectional preliminary report. BMC Med. 2011 Mar 7;9:22. doi: 10.1186/1741-7015-9-22. PMID 21385345